CLINICAL TRIAL: NCT00399256
Title: Improved Estimation of Glomerular Filtration Rate by Serum Cystatin C in Preventing Contrast Induced Nephropathy by N-Acetylcysteine or Zinc
Brief Title: Improved Estimation of GFR by Cystatin C in Preventing Contrast Induced Nephropathy by NAC or Zn
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IKP201
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Kidney Failure
Keywords: contrast-induced nephropathy; Acetylcysteine; Zinc; Cystatin C; Creatinine
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Acetylcysteine; Zinc

INTERVENTIONS:
Drug: Acetylcysteine
Drug: Zinc

SUMMARY:
Background Prevention of contrast media (CM) induced nephropathy (CIN) by pharmacological prophylaxis (e.g. N-acetylcysteine; NAC) is controversially discussed. So far, in all interventional studies assessment of kidney function was based on measurements of serum creatinine although this surrogate biomarker has several limitations. We investigated the antioxidants NAC and zinc (Zn) for the prevention of CIN by monitoring concomitantly serum levels of creatinine and cystatin C.

DETAILED DESCRIPTION:
In a prospective, placebo-controlled, double blind trial patients with moderate impaired kidney function receiving hypoosmolar, nonionic contrast medium were randomly assigned to an oral treatment for 2 days with 1.2g/day of NAC (n=19), for 1 day with 60mg/day of Zn (n=18) or placebo (n=17). All patients were periprocedural hydrated with 1ml/kg/h of 0.45% saline for 24h. At baseline (before hydration), prior to exposure of CM as well as 2 and 6 days after CM serum levels of creatinine and cystatin C have been measured.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years of age,
2. serum creatinine > 1.2 mg/dl or a creatinine clearance < 50 ml/min (measured by a 12 or 24 hour urine collection).

Exclusion Criteria:

1. acute inflammatory disease,
2. medication with NSAID or metformin until 3 days before entering study,
3. abnormal findings in physical examinations, e.g. signs of dehydration or decompensated heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Incidence of acute renal failure

SECONDARY OUTCOMES:
Rise in creatinine of > 0.5 mg/dl
Rise in creatinine > 25%
Significant rise in serum cystatin C)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik M Alscher, MD, Principal Investigator — Robert-Bosch-Hospital, Stuttgart, Germany
Locations (1):
- Robert-Bosch-Hospital, Stuttgart, Germany

REFERENCES:
- [Derived] Schanz M, Schaaf L, Dippon J, Biegger D, Fritz P, Alscher MD, Kimmel M. Renal effects of metallothionein induction by zinc in vitro and in vivo. BMC Nephrol. 2017 Mar 16;18(1):91. doi: 10.1186/s12882-017-0503-z. PMID 28302075